CLINICAL TRIAL: NCT07394933
Title: Guided Bone Regeneration Using Ti-Reinforced PTFE Membrane Vs. Khoury's Technique in Augmentation of Posterior Mandibular Defects: A Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, ahmed hassan zaher, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-019
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Atrophic Ridge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Khoury's bone shell technique (Active Comparator): Bone blocks will be harvested from the retromolar area after measuring of the size required and measuring of the donor site anatomy. Piezoelectric device will be used to perform the graft osteotomy. The block size should be slightly larger than the defect size. Sharp bony edges will be smoothened, and the donor defect will be packed with gelatin sponges. The bone block margins will be smoothened and separated into two thinner bone shells using titanium disk with copious saline irrigation. The blocks will be fixed into the recipient site buccally using at least two micro-screws leaving a gap to be filled with bone graft.
  Interventions: Procedure: Khoury's bone shell technique
- GBR using Ti-reinforced PTFE Membrane (Experimental): A non-resorbable ti-enforced polytetrafluoroethylene (PTFE) membrane will be fixed with titanium screws on the lingual bone plate and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft).
  Interventions: Procedure: GBR using Ti-reinforced PTFE Membrane

INTERVENTIONS:
Procedure: Khoury's bone shell technique — Bone blocks will be harvested from the retromolar area after measuring of the size required and measuring of the donor site anatomy. Piezoelectric device will be used to perform the graft osteotomy. The block size should be slightly larger than the defect size. Sharp bony edges will be smoothened, and the donor defect will be packed with gelatin sponges. The bone block margins will be smoothened and separated into two thinner bone shells using titanium disk with copious saline irrigation. The blocks will be fixed into the recipient site buccally using at least two micro-screws leaving a gap to be filled with bone graft.
  Arms: Khoury's bone shell technique
Procedure: GBR using Ti-reinforced PTFE Membrane — A non-resorbable ti-enforced polytetrafluoroethylene (PTFE) membrane will be fixed with titanium screws on the lingual bone plate and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft).
  Arms: GBR using Ti-reinforced PTFE Membrane

SUMMARY:
The aim of the present clinical trial is to compare two different alveolar ridge bone augmentation techniques for mandibular horizontal bone defects.

DETAILED DESCRIPTION:
Will using PTFE membrane with a mixture of xenograft and particulate autogenous bone result in bone gain similar to standard Khoury's bone shell technique?

ELIGIBILITY:
Inclusion Criteria:

1. Have one or more missing teeth in the posterior mandibular segment.
2. The alveolar ridge in the edentulous site of the selected patients will have a buccolingual width of less than 5 mm.
3. Sufficient vertical bone height above inferior alveolar nerve.
4. Free of any local or systemic condition that may contraindicate ridge expansion procedure.
5. No sex predilection.
6. The patient will be between the ages of 18-70 years.

Exclusion Criteria:

1. Patients taking any medication that may interfere with bone healing or bone biology.
2. Patients with any systemic disease that may affect bone healing.
3. Any patients with any previous bone grafting procedure at the site of interest.
4. Heavy Smokers (more than 20 cigarettes daily).
5. Patient's that have been diagnosed with periodontal disease, as sufficient ridge height would be improbable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cone Beam Volumetric Topography (CBVT) | 6 Months

SECONDARY OUTCOMES:
Clinical measurement: the frequency of complications | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - The British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided